CLINICAL TRIAL: NCT02794246
Title: Phase 2 Study Of Autologous T Cells Engineered To Express an Anti-CD19 Chimeric Antigen Receptor (CART-19) Following First-line Autologous Stem Cell Transplantation for High-risk Multiple Myeloma
Brief Title: CART-19 Post-ASCT for Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to administrative reasons.
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 19416, 824655
Record Dates: First submitted 2016-06-06; First posted 2016-06-09 (Estimated); Results first posted 2020-03-04 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental)
  Interventions: Biological: CART-19 cells

INTERVENTIONS:
Biological: CART-19 cells

SUMMARY:
This will be a single-arm, open-label study. Patients will be enrolled during induction therapy for multiple myeloma, prior to standard-of-care consolidation with autologous stem cell transplantation (ASCT). T cells will be harvested for T cell manufacturing prior to ASCT, and CART-19 will be infused at day ~60 post-ASCT, 3 days after lymphodepleting chemotherapy. The primary endpoint is progression-free survival (PFS) after ASCT. As detailed below, the study is powered to detect an increase in two-year PFS to ~75% from a baseline expectation of 55% based on historical data. Secondary endpoints will evaluate CART-19 persistence and function, minimal residual disease, immune correlative endpoints, and associations of progression-free survival (PFS) with CART-19 persistence and clinical and biologic characteristics of multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be age 18-70, inclusive, at time of enrollment.
* Subjects must have ECOG performance status of 0-2.
* Subjects must have a confirmed diagnosis of active multiple myeloma according to IMWG criteria, summarized below in Table 6. For circumstances not encompassed by this summary of the diagnostic criteria, reference can be made to the full publication of the IMWG criteria67. In addition, subjects must have "high-risk" multiple myeloma according to one of the following criteria:

  1. Any of the following high-risk cytogenetic features, documented by FISH or metaphase karyotyping: deletion 17p, t(4;14), t(14;16), t(14;20).
  2. Standard-risk cytogenetics but elevated LDH and beta-2-microglobulin > 5.5 mg/L (i.e., R-ISS stage III).
* At time of enrollment, subjects must be within 9 months of initiation of systemic therapy for multiple myeloma.
* Requirements for pre-enrollment therapy: Subjects must have received or be receiving, at time of enrollment, "RVD" therapy (combination therapy with lenalidomide, bortezomib, and dexamethasone). Patients must have received ≤6 cycles of RVD at time of enrollment and must not have progressed (by IMWG criteria65) on RVD. Patients may have received other regimens prior to RVD if such therapy was limited to ≤3 cycles. Patients may have received radiation therapy prior to enrollment. Patients must not have received infusional chemotherapy (e.g., VTD-PACE or similar regimen) prior to enrollment.
* Subjects must be eligible for ASCT and to receive a melphalan dose of 200 mg/m2 as defined by the following criteria:

  1. Left ventricular ejection fraction ≥ 40%,
  2. AST/ALT ≤2.5 times the upper limit of normal
  3. Total bilirubin ≤1.5 mg/dL, unless hyperbilirubinemia is attributable solely to Gilbert's syndrome.
  4. Estimated (by CKD-EPI or Cockgroft-Gault equations) or calculated CrCl ≥40 ml/min.
  5. DLCO ≥50% of predicted after correction for anemia.
* Subjects must have measurable disease by standard serum and urine tests to enable post-transplant monitoring for progression-free survival. Any of the following criteria are sufficient to define measurable disease.

  1. Serum M-spike ≥ 0.5 g/dL
  2. 24 hr urine M-spike ≥ 200mg
  3. Involved serum FLC ≥ 50 mg/L with abnormal ratio
  4. For IgA multiple myeloma, total serum IgA level elevated above normal range. Note: Measurable disease does not need to be documented at enrollment but can be based on historical lab results obtained at or since diagnosis with multiple myeloma. For example, a patient who does not have measurable disease at enrollment due to complete remission after induction therapy is eligible if the disease was previously measurable by one of the above criteria.
* Subjects must have signed written, informed consent.
* Subjects of reproductive potential must agree to use acceptable birth control methods

Exclusion Criteria:

* Subjects must not:

Be pregnant or lactating. Have inadequate venous access for or contraindications to leukapheresis. Have any active and uncontrolled infection. Any uncontrolled medical or psychiatric disorder that would preclude participation as outlined.

Have NYHA Class III or IV heart failure (see Appendix 2), unstable angina, or a history of recent (within 6 months) myocardial infarction or sustained (>30 seconds) ventricular tachyarrhythmias.

Have undergone allogeneic stem cell transplantation. Have received prior gene therapy or gene-modified cellular immunotherapy. Have active auto-immune disease, including connective tissue disease, uveitis, sarcoidosis, inflammatory bowel disease, or multiple sclerosis, or have a history of severe (as judged by the principal investigator) autoimmune disease requiring prolonged immunosuppressive therapy.

Have prior or active central nervous system (CNS) involvement (e.g. leptomeningeal disease, parenchymal masses) with myeloma. Screening for this (e.g. with lumbar puncture) is not required unless suspicious symptoms are present.

Have a contraindication to post-ASCT maintenance lenalidomide. Have active infection with HIV (negative HIV 1/2 antibody screen), hepatitis C (negative hepatitis C antibody screen), or hepatitis B (negative hepatitis B surface antigen). Any positive serologies for HIV or viral hepatitis should be confirmed with appropriate confirmatory testing before concluding that an active infection is present. Subjects with positive hepatitis core antibody are also excluded since the effect of long-term B cell depletion on the risk of hepatitis B reactivation is unknown.

Patients with a known history or prior diagnosis of optic neuritis or other immunologic or inflammatory disease affecting the central nervous system.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alfred Garfall, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- CART-19 Cells: single infusion of 1-5x10E8 cells CART-19 cells
Period: Overall Study
Arm/Group | CART-19 Cells
Started | 6
Treated | 3
Completed | 0
Not Completed | 6
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 4

BASELINE CHARACTERISTICS:
Groups:
- Single Arm: CART-19 cells
Arm/Group | Single Arm
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Evaluate Progression Free Survival
Description: Progression free survival as defined by Partial Response (PR); Stable Disease (SD); Very Good Partial Response (VGPR), and Stringent Complete Response (sCR) to treatment. The outcome measures range from Stable disease to Stringent Complete Response (SD worst outcome; sCR best outcome
Time Frame: Follow progression-free survival (PFS) for 2-3 years post CART-19 infusion
Measure: Number; unit: participants
Arm/Group | Single Arm
Number analyzed (Participants) | 6
participants
  Stable Disease | 1
  Partial Response | 3
  Very Good Partial Response | 1
  Stringent Complete Response | 1

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=6)
Upper respiratory infection (Infections and infestations) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=6)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 1 (1) — non-serious grade 2 AE
Platelet count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-04-11): https://cdn.clinicaltrials.gov/large-docs/46/NCT02794246/Prot_SAP_000.pdf
  • Informed Consent Form (2017-04-11): https://cdn.clinicaltrials.gov/large-docs/46/NCT02794246/ICF_001.pdf